CLINICAL TRIAL: NCT04731220
Title: A Questionnaire Survey Study for Establishment of Surveillance and Prevention Through the Analysis of Epidemiologic Risk Factors in Patients With Biliary Tract Cancers
Brief Title: A Questionnaire Survey for Biliary Tract Cancers
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Kyungpook National University Chilgok Hospital (Other)
Collaborators: Kyungpook National University Hospital (Other); Pusan National University Hospital (Other); Pusan National University Yangsan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KNUCH 2020-04-045
Record Dates: First submitted 2021-01-20; First posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Newly diagnosed as bile duct cancer
- Control group: No history of cancer in previous 5 years

SUMMARY:
The purpose of this study is:

* To evaluate risk factors for cancers of the biliary tract by registering new patients and their counterparts in a multi-center program
* Development of programs by creating a multi-center biliary tract cancer registration system

ELIGIBILITY:
Inclusion Criteria:

* Study population :

  * Newly diagnosis of biliary tract cancers - Pathological or Radiological or other clinical diagnosis of biliary tract cancers
  * Informed consent
* Control :

  * with no previous cancer diagnosis
  * Informed consent

Exclusion Criteria:

* Previous diagnosis of bile duct cancer with resection operation, endoscopic resection, chemotherapy or radiation therapy
* Prior diagnosis of other cancer in 5 years or ongoing cancer treatment
* Patients' refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population should be defined in advance, stating eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of cases and controls who complete each part of the study | 5 years
  Information is obtained by a questionnaire, laboratory findings, image data, physiological parameter.

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook National University Chilgok Hospital, Daegu, South Korea